CLINICAL TRIAL: NCT03612817
Title: A 3-month Study Investigating the 24-hour Efficacy With the Preservative-free Tafluprost/Timolol Fixed Combination Dosed Morning, or Evening in Subjects With Open-angle Glaucoma Insufficiently Controlled With Latanoprost Monotherapy
Brief Title: Preservative-free Tafluprost/Timolol Fixed Combination: Morning vs Evening Dosing
Acronym: TTFC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Santen Oy (Industry)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 433
Record Dates: First submitted 2018-07-20; First posted 2018-08-02 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Glaucoma, Open-Angle
Keywords: tafluprost/timolol fixed combination, 24-hour IOP control
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — tafluprost

STUDY DESIGN:
Intervention Model Description: Patients first undergo a baseline, habitual 24-hour pressure assessment with branded, or generic latanoprost. Suitably qualified open-angle glaucoma patients (latanoprost-treated, mean 24-hour pressure greater than 20 mm Hg) are randomized for Period 1 to receive either tafluprost/timolol fixed combination drops once in the evening (20:00) and placebo drops in the morning (08:00), or tafluporst/timolol drops once in the morning (08:00) and placebo in the evening (20:00). After 3 months of chronic therapy (± 2 weeks) study patients undergo a treated, habitual 24-hour pressure assessment. Study subjects are then switched to the opposite treatment regimen for Period 2 (tafluprost/timolol in the evening instead of morning etc) and after another 3 months they undergo the third and final evaluation of their 24-hour pressure.
Who Masked: Investigator
Masking Description: Only the dosing coordinator is aware of the treatment used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tafluprost/timolol with PM dosing (Active Comparator): Therapy with Tafluprost/timolol fixed combination drops dosed PM (20:00)
  Interventions: Drug: Tafluprost/timolol fixed combination
- Tafluprost/timolol with AM dosing (Active Comparator): Therapy with Tafluprost/timolol fixed combination drops dosed AM (08:00)
  Interventions: Drug: Tafluprost/timolol fixed combination

INTERVENTIONS:
Drug: Tafluprost/timolol fixed combination — Evaluation of 24-hour pressure control with tafluprost/timolol given in the evening or morning
  Other Names: Taptiqom

SUMMARY:
The ideal dosing for preservative-free tafluprost/timolol fixed combination remains to be elucidated. The present study compared the 24-hour intraocular pressure efficacy obtained with tafluprost/timolol given once in the evening with placebo once in the morning, versus that with the same fixed combination administered once in the morning with placebo given once in the evening in consecutive patients with open-angle glaucoma insufficiently controlled with branded, or generic latanoprost monotherapy.

DETAILED DESCRIPTION:
Prospective, observer-masked, placebo-controlled, crossover, comparison in consecutive open-angle glaucoma patients, insufficiently controlled with preserved latanoprost monotherapy (mean 24-hr IOP greater than 20 mmHg). Patients were randomized to either morning (08:00), or evening (20:00) preservative-free tafluprost/timolol fixed combination for 3 months and then were crossed over. After each treatment period patients underwent habitual 24-hour intraocular pressure monitoring with Goldmann tonometry in the sitting position (at 10:00, 14:00, 18:00 and 22:00) and Perkins tonometry in the supine position (at 02:00 and 06:00).

Primary Study Objective: Mean 24-hour efficacy with both dosing regimens of tafluprost/timolol fixed combination versus latanoprost monotherapy.

Secondary Study Objectives

1. Mean efficacy with the evening dosing of tafluprost/timolol compared with the morning-dosed tafluprost/timolol fixed combination at each time point measured.
2. Mean daytime and mean nighttime IOP control with the two dosing regimens.
3. Mean peak and fluctuation of 24-hour pressure with the evening and the morning dosing of the fixed combination.

ELIGIBILITY:
Inclusion Criteria:

1. age between 21-85 years;
2. mild to moderate glaucomatous disc damage and visual field loss (less than -12 dB mean deviation visual field loss attributed to glaucoma and 0.8 or better vertical cup-to-disc ratio);
3. visual acuity greater than 0.1 in the study eye;
4. open anterior chamber angles;
5. in each patient the diagnosis of open-angle glaucoma will be made by the principal investigator based on the European Glaucoma Society criteria;
6. study patients will have to demonstrate a reliable visual field (at least two visual fields with less than 20% fixation losses, false positives, or negatives);
7. patient should understand the study instructions and to be willing to attend all follow-up appointments and should be willing to comply with study medication usage.

Exclusion Criteria:

1. previous history of less than 10% IOP decrease on any IOP-lowering medication;
2. evidence of concurrent conjunctivitis, keratitis, or uveitis in either eye;
3. history of inadequate adherence; intolerance, or contraindication to either prostaglandins, β-blockers, dorzolamide, or benzalconium chloride (BAK);
4. severe ocular surface disease, intraocular conventional or laser surgery in the study eye (within 6 months prior to enrolment);
5. previous history of ocular trauma;
6. use of corticosteroids (within 3 months before the enrolment) and use of contact lenses;
7. patients will also be excluded if on baseline exam they show clinical evidence of inflammation, signs of ocular infection (except blepharitis), signs of any corneal abnormality that will affect subsequent IOP measurements;
8. unwillingness to participate in the trial;
9. females of childbearing potential or lactating mothers.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Mean 24-hour pressure control with Tafluprost/timolol fixed combination dosed morning or evening | 3-month study
  24-hour efficacy documented after each period of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Giannopoulos, MD, Study Director — Aristotle University
Locations (1):
- 1st University Department of Ophthalmology, Thessaloniki, Makedonia, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Konstas AG, Katsanos A, Athanasopoulos GP, Voudouragkaki IC, Panagiotou ES, Pagkalidou E, Haidich AB, Giannoulis DA, Spathi E, Giannopoulos T, Katz LJ. Preservative-free tafluprost/timolol fixed combination: comparative 24-h efficacy administered morning or evening in open-angle glaucoma patients. Expert Opin Pharmacother. 2018 Dec;19(18):1981-1988. doi: 10.1080/14656566.2018.1534958. Epub 2018 Oct 17. PMID 30328725